CLINICAL TRIAL: NCT05533502
Title: Acute Effects of a Combination Plant-Based Protein and Marine-Based Multi-Mineral Supplement on Postprandial Gut Hormones and Bone Remodeling in Young Adults
Brief Title: Combination Plant-Based Protein and Marine-Based Multi-Mineral Supplement and Bone Remodeling in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: Marigot Ltd. (Industry); Enterprise Ireland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2022_03_06_EHS
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2022-09

CONDITIONS: Bone Resorption; Bone and Bones
Keywords: nutrition; plant; marine; protein; bone; skeletal; health; dietary supplements; sustainable
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Intervention Model Description: A block-randomized, within-subject, two-day, crossover design examining acute (0-4 h) postprandial changes in different gut hormone concentrations and bone remodeling biomarkers in 12 healthy, young adults following ingestion of a combination plant-based protein and marine-based multi-mineral supplement or control.
Who Masked: Investigator
Masking Description: Single Blind Study (Investigator only)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Supplement: Combined Plant-Based Protein and Marine-Based Multi-Mineral Supplement (Active Comparator): Fava-Bean Protein Concentrate and Aquamin F
  Interventions: Dietary Supplement: Combined Plant-Based Protein and Marine-Based Multi-Mineral Supplement
- Placebo Control (Placebo Comparator): Placebo Control
  Interventions: Dietary Supplement: Placebo Control

INTERVENTIONS:
Dietary Supplement: Combined Plant-Based Protein and Marine-Based Multi-Mineral Supplement — Ingestion of the Test Product at 07.00am - Fava-bean protein concentrate dosed at 0.33 g/kg body mass and Aquamin F dosed at 800mg in 500 ml water volume. Supplied by Marigot Limited, Strand Farm Currabinny, Co. Cork, Ireland
  Arms: Dietary Supplement: Combined Plant-Based Protein and Marine-Based Multi-Mineral Supplement
Dietary Supplement: Placebo Control — Ingestion of the Control Product at 07.00am - 500ml water volume.
  Arms: Placebo Control

SUMMARY:
Nutrient intake of calcium and protein are known to function as regulators of bone remodeling. Specifically, a balanced rate of bone resorption and bone formation (i.e. bone remodeling process) is required to maintain bone health. However, a high remodeling rate, or an imbalance between formation and resorption, as well as suboptimal nutrient intake are known to contribute to fracture risk and bone dysfunction.

Gut-derived hormones represent an important link between nutrient intake and bone remodeling (i.e. gut-bone axis). A sustainable nutritional intervention that positively modulates the postprandial responses of gut-derived hormones and the linked bone remodeling processes is an attractive option for the optimization of bone health in young adults.

The proposed nutrient intervention seeks to explore the bioefficacy of a combination plant-based protein and marine-based multi-mineral supplement following oral ingestion in young, healthy men and women. A postprandial time-course study will be undertaken to examine the acute effects and/or associations between different gut-derived hormones and biomarkers of bone metabolism.

DETAILED DESCRIPTION:
A block-randomized, within-subject, two-day, crossover design examining acute (0-4 hour) postprandial changes in different gut-derived hormone concentrations and biomarkers of bone metabolism in 12 healthy, young adults following ingestion of a combination plant-based protein and marine-based multi-mineral supplement or control.

Each participant will consume (in a random manner) either one of two investigational products (i.e., combined nutritional supplement or control). The combined nutritional supplement will consist of: 0.3 g/kg body mass of ATURA Fava-Bean Protein and 800mg of Aquamin F (a highly bioactive source of minerals rich in calcium) dissolved in 500ml water volume. The control product will consist of 500ml water volume without the protein and multi-mineral nutritional composition.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 35 years.
* Recreationally active (150-300 min/week of moderate physical activity).
* Healthy (i.e.,not presenting with injury, illness, medication, history of chronic disease, or known allergies/intolerance (e.g. favism) to the ingredients contained in either formulation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Bone turnover | Pre-ingestion and 15, 30, 45, 60, 90, 120, 180, 240 minutes Post-ingestion (Plasma)
  A balance of the difference between the magnitude and time course of the acute change (0-4 hours) in plasma C-terminal telopeptide of type 1 collagen (CTX) in ng/mL, a measure of bone resorption, and procollagen type 1 amino-terminal propeptide (P1NP) in ng/ml, a measure of bone formation.

SECONDARY OUTCOMES:
Change in regulator of bone metabolism - Parathyroid hormone | Pre-ingestion and 15, 30, 45, 60, 90, 120, 180, 240 minutes Post-ingestion (Plasma)
  The magnitude and time course of the acute change (0-4 hours) in plasma parathyroid hormone (PTH) measured in pmol/L.
Change in ionized calcium and potassium. | Pre-ingestion and 15, 30, 45, 60, 90, 120, 180, 240 minutes Post-ingestion (Whole Blood)
  The magnitude and time course of the acute change (0-4 hours) in ionized calcium and potassium.
Vitamin D Status | Pre-ingestion (Plasma)
  Pre-ingestion total plasma 25 (OH)D level
Change in insulin and glucose | Pre-ingestion and 15, 30, 45, 60, 90, 120, 180, 240 minutes Post-ingestion (Plasma)
  The magnitude and time course of the acute change (0-4 hours) in plasma insulin and glucose
Change in incretin peptides | Pre-ingestion and 15, 30, 45, 60, 90, 120, 180, 240 minutes Post-ingestion (Plasma)
  The magnitude and time course of the acute change (0-4 hours) in enterogastric peptide glucose-dependent insulinotropic peptide (GIP1-42) measured in pg/mL, glucagon-like peptide-1 (GLP-17-36) measured in pg/mL and GLP-2 (1-33) measured in pg/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Jakeman, PhD, Principal Investigator — University of Limerick
Locations (1):
- Faculty of Education & Health Sciences, University of Limerick,, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://aquamin.com/products/marine-minerals-aquamin-f/
- See also: Related Info — https://aturaproteins.com/plant-proteins/fava-bean-protein/